CLINICAL TRIAL: NCT02642471
Title: Sentinel Lymph Node Biopsy Versus Pelvic Lymphadenectomy in Early-stage Cervical Cancer (PHENIX/CSEM 010)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jihong Liu, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-FXY-073
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer; Surgery; Quality of Life
Keywords: sentinel lymph node; pelvic lymphadenectomy; cervical carcinoma; surgery; radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Experimental): patients with negative sentinel nodes confirmed by pathological examination of frozen section will be randomly assigned to Arm 1 or Arm 2 Arm 1: patients undergo radical hysterectomy±salpingo-oophorectomy (no systematic pelvic lymphadenectomy) Arm 2: patients undergo radical hysterectomy±salpingo-oophorectomy+pelvic lymph node dissection
  Interventions: Procedure: no systematic pelvic lymphadenectomy
- Arm 2 (No Intervention): patients with negative sentinel nodes confirmed by pathological examination of frozen section will be randomly assigned to Arm 1 or Arm 2 Arm 1: patients undergo radical hysterectomy±salpingo-oophorectomy (no systematic pelvic lymphadenectomy) Arm 2: patients undergo radical hysterectomy±salpingo-oophorectomy+pelvic lymph node dissection
- Arm 3 (Experimental): patients with positive sentinel nodes confirmed by pathological examination of frozen section will be randomly assigned to Arm 3 or Arm 4 Arm 3: patients undergo radical hysterectomy±salpingo-oophorectomy (no systematic pelvic lymphadenectomy) Arm 4: patients undergo radical hysterectomy±salpingo-oophorectomy+pelvic lymph node dissection
  Interventions: Procedure: no systematic pelvic lymphadenectomy
- Arm 4 (No Intervention): patients with positive sentinel nodes confirmed by pathological examination of frozen section will be randomly assigned to Arm 3 or Arm 4 Arm 3: patients undergo radical hysterectomy±salpingo-oophorectomy (no systematic pelvic lymphadenectomy) Arm 4: patients undergo radical hysterectomy±salpingo-oophorectomy+pelvic lymph node dissection

INTERVENTIONS:
Procedure: no systematic pelvic lymphadenectomy — systematic pelvic lymphadenectomy is omitted in surgical treatment
  Arms: Arm 1; Arm 3

SUMMARY:
The diagnostic value of sentinel lymph node biopsy in early-stage cervical cancer has been well studied. However, there were no randomized controlled study on comparing the long-term outcomes of sentinel lymph node biopsy and conventional procedure. The investigators perform a phase III, randomized controlled trial to determine whether pelvic lymphadenectomy can be replaced by sentinel lymph node biopsy in surgical treatment for patients with early-stage cervical cancer.

DETAILED DESCRIPTION:
This study comprises two parts: PHENIX-I: To compare the outcomes of managements with and without pelvic lymphadenectomy for patients with negative sentinel lymph node; PHENIX-II: To compare the outcomes of managements with and without pelvic lymphadenectomy for patients with positive sentinel lymph node. Patients with newly diagnosed International Federation of Gynecology and Obstetrics (FIGO) stage IA1 (lymphovascular space involvement), IA2, IB1, and IB2 cervical cancer are eligible for our study. The tumor diameter should be less than 3cm. Sentinel lymph node biopsy will be performed at the beginning of operations. After pathological examination of frozen section, patients will be assigned to PHENIX-I or PHENIX-II study according to their status of sentinel nodes. In both parts of this trail, patients have equal chance to be randomly assigned to experimental arms (radical hysterectomy only) and reference arms (radical hysterectomy and pelvic lymphadenectomy).Adjuvant treatments will be planned according to postoperative pathological factors. The primary objective is disease-free survival at 3 years for PHENIX-I and 2 years for PHENIX-II. The secondary end points are overall survival, long-term outcome of sentinel lymph node biopsy and the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed cervical carcinoma
* Histopathology squamous carcinoma, adenocarcinoma or adeno-squamous carcinoma
* Original clinical stage must be FIGO (2018) stage IA1 (lymphovascular space involvement), IA2, IB1, IB2 and IIA1
* No suspected node should be found on imaging examination (RESIST 1.1)
* Age between 18-65
* Patients must give signed informed consent
* P.S status: 0-1
* Estimated survival time > 3 months
* Tumor diameter ≤ 3 cm

Exclusion Criteria:

* The presence of uncontrolled life-threatening illness
* Receiving other ways of anti-cancer therapy
* Investigator consider the patients can't finish the whole study
* With normal liver function test (ALT、AST>2.5×ULN)
* With normal renal function test (Creatinine>1.5×ULN)
* WBC<4,000/mm3 or PLT<100,000/mm
* The whole cervix has been occupied by tumor and there is no normal surface left for tracer injection
* History of severe heart disease or deep venous thrombosis; 4) Presence or history of other malignant disease
* Gestation or perinatal period
* Intention to fertility preservation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2015-12-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival in PHENIX-I | 3 years
Disease free survival in PHENIX-II | 2 years

SECONDARY OUTCOMES:
Surgical morbidity | 3 years
Rate of retroperitoneal node recurrence | 3 years
Overall survival | 5 years
Patients' quality of life | 5 years
Performance of SLN detection | 3 years
Diagnostic accuracy of frozen section examination | 3 years
Anatomic distribution of SLNs | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Ph. D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Gynecologic Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tu H, Huang H, Li Y, Chen X, Wang C, Zheng M, Zhang Y, Zhao W, Feng Y, Wan T, Huang Y, Yu A, Lu W, Xiao J, Shan W, Zhang P, Zhu C, Wang D, Zhou H, Li J, Kong B, Feng W, Wang X, Luo R, Huang X, Li J, Lin Z, Yao S, Liu J; PHENIX Investigators. Sentinel-Lymph-Node Biopsy Alone or with Lymphadenectomy in Cervical Cancer. N Engl J Med. 2025 Oct 16;393(15):1463-1474. doi: 10.1056/NEJMoa2506267. PMID 41092328
- [Derived] Tu H, Huang H, Xian B, Li J, Wang P, Zhao W, Chen X, Xie X, Wang C, Kong B, Xiao J, Zhang P, Liu J; PHENIX Investigators and the CSEM group. Sentinel lymph node biopsy versus pelvic lymphadenectomy in early-stage cervical cancer: a multi-center randomized trial (PHENIX/CSEM 010). Int J Gynecol Cancer. 2020 Nov;30(11):1829-1833. doi: 10.1136/ijgc-2020-001857. Epub 2020 Sep 24. PMID 32973117